CLINICAL TRIAL: NCT05438134
Title: Enhancing Resilience in Senior Living Community Residents: A Randomized Controlled Trial
Brief Title: Enhancing Resilience in Senior Community Residents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Lara Traeger, Assistant Professor, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2021A019096
Record Dates: First submitted 2022-06-24; First posted 2022-06-29 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-11

CONDITIONS: Quality of Life; Stress, Psychological
Keywords: Resiliency; Flourishing; Coping Skills; Stress Reduction; Healthy Aging
MeSH Terms: conditions — Stress, Psychological

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SMART-3RP Group Intervention (Experimental): Residents will participate in 9 structured weekly group sessions which incorporates stress management and relaxation training upon enrollment.
  Interventions: Behavioral: SMART-3RP Group Intervention
- Waitlist Control Group Intervention (Active Comparator): Residents will participate in 9 structured weekly group sessions which incorporates stress management and relaxation training after the final survey time point.
  Interventions: Behavioral: SMART-3RP Group Intervention

INTERVENTIONS:
Behavioral: SMART-3RP Group Intervention — Nine 1.5 hour group sessions focusing on developing:
  1. An understanding of stress physiology and the physiology of the relaxation response;
  2. A regular practice of eliciting the relaxation response; and
  3. Cognitive behavioral and positive psychology/resilience skills.
  Participants receive a copy of the SMART-3RP session manual and audio recorded guided meditations for independent relaxation practice. Participants are encouraged to practice eliciting the relaxation response daily throughout the study, using the audio recordings or other mind body techniques. Participants will use a practice log to track their practice.

SUMMARY:
This randomized waitlist-controlled trial tests the efficacy of the Stress Management and Resiliency Training Relaxation Response Resiliency Program (SMART-3RP), a mind-body intervention, to enhance resilience and flourishing among residents in continuing care retirement communities. The investigators hypothesize that participants in the SMART-3RP group will report greater increases in resilience and flourishing relative to participants in the control group.

DETAILED DESCRIPTION:
This randomized control trial tests the efficacy of the Stress Management and Resiliency Training Relaxation Response Resiliency Program (SMART-3RP) to improve resilience and flourishing among older adults residing in continuing care retirement communities relative to a wait-list control group. At enrollment, participants will be randomly assigned to the intervention group or the control group using computer generated 1:1 blocked randomization stratified by community site. The intervention group will receive the SMART-3RP program immediately upon enrollment; the wait-list control group will be invited to receive the SMART-3RP program after the final survey time point. An estimate of 360 participants will be recruited from up to nine geographically diverse Erickson Senior Living communities.

ELIGIBILITY:
Inclusion Criteria:

* Resident of an Erickson Senior Living community
* Currently residing in an Erickson Senior Living apartment home
* Sufficient English language skills to participate in study procedures

Exclusion Criteria:

* Unable or unwilling to provide informed consent
* Unable or unwilling to participate in in-person group sessions

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 288 (Actual)
Dates: Start 2022-06-24 (Actual); Primary Completion 2023-04-05 (Actual); Study Completion 2023-04-05 (Actual)

PRIMARY OUTCOMES:
Resilience: Current Experiences Scale (CES) | Up to 12 weeks
  We will investigate longitudinal differences in resilience between study groups (CES score range 0-115), with higher scores indicating greater resilience.
Flourishing: Flourishing Measure (FM) | Up to 12 weeks
  We will investigate longitudinal differences in flourishing between study groups (FM score range 0-10), with higher scores indicating greater flourishing.

SECONDARY OUTCOMES:
Psychological distress: Patient Health Questionnaire 4 (PHQ4) | Up to 12 weeks
  We will investigate longitudinal differences in psychological distress between study groups (PHQ4 score range 0-12), with higher scores indicating greater distress.
Social isolation: Patient-Reported Outcomes Measurement Information System - Social Isolation (PROMIS-SI) | Up to 12 weeks
  We will investigate longitudinal differences in social isolation between study groups (PROMIS-SI score range 4-20), with higher scores indicating greater isolation.
Physical symptoms: Condensed Memorial Symptom Assessment Scale (CMSAS) | Up to 12 weeks
  We will investigate longitudinal differences in physical symptom burden between study groups (CMSAS score range 0-48, with higher scores indicating greater symptom burden.
Coping self-efficacy: Measure of Current Status - Part A (MOCS-A) | Up to 12 weeks
  We will investigate longitudinal differences in coping self-efficacy between study groups (MOCS-A score range 0-52), with higher scores indicating greater self-efficacy.
Community well-being: Community Well Being Survey (CWB) | Up to 12 weeks
  We will investigate longitudinal differences in community well-being between study groups (CWB range 0-10), with higher scores indicating greater community well-being.
Positive affect: Positive and Negative Affect Schedule - Positive Subscale (PANAS-POS) | Up to 12 weeks
  We will investigate longitudinal differences in positive affect between study groups (PANAS-POS range 10-50), with higher scores indicating greater positive affect.

CONTACTS AND LOCATIONS:
Overall Officials: Lara Traeger, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Background] McEwen BS, Stellar E. Stress and the individual. Mechanisms leading to disease. Arch Intern Med. 1993 Sep 27;153(18):2093-101. PMID 8379800
- [Background] UN Dept of Economic and Social Affairs, Population Division. Population ageing and development: ten years after Madrid. Population Facts. 2012;No. 2012/4.
- [Background] Park ER, Traeger L, Vranceanu AM, Scult M, Lerner JA, Benson H, Denninger J, Fricchione GL. The development of a patient-centered program based on the relaxation response: the Relaxation Response Resiliency Program (3RP). Psychosomatics. 2013 Mar-Apr;54(2):165-74. doi: 10.1016/j.psym.2012.09.001. Epub 2013 Jan 22. PMID 23352048
- [Background] VanderWeele TJ. On the promotion of human flourishing. Proc Natl Acad Sci U S A. 2017 Aug 1;114(31):8148-8156. doi: 10.1073/pnas.1702996114. Epub 2017 Jul 13. PMID 28705870
- [Background] Park ER, Perez GK, Millstein RA, Luberto CM, Traeger L, Proszynski J, Chad-Friedman E, Kuhlthau KA. A Virtual Resiliency Intervention Promoting Resiliency for Parents of Children with Learning and Attentional Disabilities: A Randomized Pilot Trial. Matern Child Health J. 2020 Jan;24(1):39-53. doi: 10.1007/s10995-019-02815-3. PMID 31650412
- [Background] Gonzalez A, Shim M, Mahaffey B, Vranceanu AM, Reffi A, Park ER. The Relaxation Response Resiliency Program (3RP) in Patients with Headache and Musculoskeletal Pain: A Retrospective Analysis of Clinical Data. Pain Manag Nurs. 2019 Feb;20(1):70-74. doi: 10.1016/j.pmn.2018.04.003. Epub 2018 Dec 13. PMID 29773354
- [Background] Vranceanu AM, Riklin E, Merker VL, Macklin EA, Park ER, Plotkin SR. Mind-body therapy via videoconferencing in patients with neurofibromatosis: An RCT. Neurology. 2016 Aug 23;87(8):806-14. doi: 10.1212/WNL.0000000000003005. Epub 2016 Jul 22. PMID 27449066
- [Background] Stahl JE, Dossett ML, LaJoie AS, Denninger JW, Mehta DH, Goldman R, Fricchione GL, Benson H. Relaxation Response and Resiliency Training and Its Effect on Healthcare Resource Utilization. PLoS One. 2015 Oct 13;10(10):e0140212. doi: 10.1371/journal.pone.0140212. eCollection 2015. PMID 26461184
- [Background] Scult M, Haime V, Jacquart J, Takahashi J, Moscowitz B, Webster A, Denninger JW, Mehta DH. A healthy aging program for older adults: effects on self-efficacy and morale. Adv Mind Body Med. 2015 Winter;29(1):26-33. PMID 25607120
- [Background] Nasreddine, Z. (2019). Montreal Cognitive Assessment FAQ, Can the MoCA be administered remotely? Retrieved from https://www.mocatest.org/faq/
- [Background] Browne RH. On the use of a pilot sample for sample size determination. Stat Med. 1995 Sep 15;14(17):1933-40. doi: 10.1002/sim.4780141709. PMID 8532986
- [Background] Lancaster GA, Dodd S, Williamson PR. Design and analysis of pilot studies: recommendations for good practice. J Eval Clin Pract. 2004 May;10(2):307-12. doi: 10.1111/j..2002.384.doc.x. PMID 15189396
- [Background] Rounsaville BJ, Carroll KM, Onken LS. A Stage Model of Behavioral Therapies Research: Getting Started and Moving on From Stage I. Clin Psychol Sci Pract. 2001;8(2):133-142. doi:https://doi.org/10.1093/clipsy.8.2.133
- [Background] Shih WJ, Ohman-Strickland PA, Lin Y. Analysis of pilot and early phase studies with small sample sizes. Stat Med. 2004 Jun 30;23(12):1827-42. doi: 10.1002/sim.1807. PMID 15195318
- [Background] Whitehead AL, Julious SA, Cooper CL, Campbell MJ. Estimating the sample size for a pilot randomised trial to minimise the overall trial sample size for the external pilot and main trial for a continuous outcome variable. Stat Methods Med Res. 2016 Jun;25(3):1057-73. doi: 10.1177/0962280215588241. Epub 2015 Jun 19. PMID 26092476
- [Background] Park ER, Luberto CM, Chad-Friedman E, Traeger L, Hall DL, Perez GK, Goshe B, Vranceanu AM, Baim M, Denninger Md PhD JW, Fricchione Md G, Benson Md H, Lechner SC. A Comprehensive Resiliency Framework: Theoretical Model, Treatment, and Evaluation. Glob Adv Health Med. 2021 Mar 24;10:21649561211000306. doi: 10.1177/21649561211000306. eCollection 2021. PMID 34377598
- [Background] Węziak-Białowolska D, McNeely E, VanderWeele T. Flourish Index and Secure Flourish Index - Development and Validation (SSRN Scholarly Paper ID 3145336). Soc Sci Res Netw. 2017.
- [Background] Antoni MH, Lechner SC, Kazi A, Wimberly SR, Sifre T, Urcuyo KR, Phillips K, Gluck S, Carver CS. How stress management improves quality of life after treatment for breast cancer. J Consult Clin Psychol. 2006 Dec;74(6):1143-52. doi: 10.1037/0022-006X.74.6.1152. PMID 17154743
- [Background] VanderWeele TJ. Measures of community well-being: A template. Int J Community Well-Being. 2019;2(3):253-275. https://doi.org/10.1007/s42413-019-00036-8
- [Background] Watson D, Clark LA, Tellegen A. Development and validation of brief measures of positive and negative affect: the PANAS scales. J Pers Soc Psychol. 1988 Jun;54(6):1063-70. doi: 10.1037//0022-3514.54.6.1063. PMID 3397865
- [Background] Hahn EA, DeWalt DA, Bode RK, Garcia SF, DeVellis RF, Correia H, Cella D; PROMIS Cooperative Group. New English and Spanish social health measures will facilitate evaluating health determinants. Health Psychol. 2014 May;33(5):490-9. doi: 10.1037/hea0000055. Epub 2014 Jan 20. PMID 24447188
- [Background] Kroenke K, Spitzer RL, Williams JB, Lowe B. An ultra-brief screening scale for anxiety and depression: the PHQ-4. Psychosomatics. 2009 Nov-Dec;50(6):613-21. doi: 10.1176/appi.psy.50.6.613. PMID 19996233
- [Background] Chang VT, Hwang SS, Feuerman M, Kasimis BS, Thaler HT. The memorial symptom assessment scale short form (MSAS-SF). Cancer. 2000 Sep 1;89(5):1162-71. doi: 10.1002/1097-0142(20000901)89:53.0.co;2-y. PMID 10964347
- [Background] Thornton M, Travis SS. Analysis of the reliability of the modified caregiver strain index. J Gerontol B Psychol Sci Soc Sci. 2003 Mar;58(2):S127-32. doi: 10.1093/geronb/58.2.s127. PMID 12646602
- [Background] Wongpakaran T, Wongpakaran N, Intachote-Sakamoto R, Boripuntakul T. The Group Cohesiveness Scale (GCS) for psychiatric inpatients. Perspect Psychiatr Care. 2013 Jan;49(1):58-64. doi: 10.1111/j.1744-6163.2012.00342.x. Epub 2012 Jun 12. PMID 23293998